CLINICAL TRIAL: NCT04332315
Title: Short and Middle Term Results of Vaginally Assisted Laparoscopic Sacropolpopexy
Brief Title: Vaginally Assisted Laparoscopic Sacropolpopexy
Acronym: VALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Aydın, Associate Prof, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VALS01
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VALS (Active Comparator): Vaginally asissted laparoscopic sacrocolpopexy
  Interventions: Procedure: Vaginally assisted laparoscopic sacrocolpopexy
- AS (Active Comparator): Abdominal Sacrocolpopexy
  Interventions: Procedure: Vaginally assisted laparoscopic sacrocolpopexy

INTERVENTIONS:
Procedure: Vaginally assisted laparoscopic sacrocolpopexy — The VALS procedure consists of two steps. First, vaginal hysterectomy or laparoscopically assisted vaginal hysterectomy performed, anterior vaginal wall dissected up to bladder neck starting from initial vaginal incision, posterior vaginal wall dissected from rectum starting from initial vaginal incision up to distal third of posterior vaginal wall.The free arms of fixed meshes are introduced to the peritoneal cavity and the vaginal vault is closed with absorbable polyglactin suture. laparoscopy phase was performed with one intraumbilical (10 mm), 3 lateral abdominal (5 mm) trocars. Two mesh strips fixated to anterior longitudinal ligament of the sacrum with two separate no: 1 polypropylene sutures without tension.
  AS was performed via Pfannenstiel incision after total or subtotal abdominal hysterectomy
  Other Names: Abdominal sacrocolpopexy

SUMMARY:
Introduction and Hypothesis: Vaginally assisted laparoscopic sacrocolpopexy (VALS), which is a combined surgical approach where a vaginal hysterectomy is initially performed, followed by transvaginal placement of synthetic mesh and laparoscopic suspension, can be an alternative to overcome the dissection, suturing limitations of laparoscopic sacrocolpopexy. The aim of this study was to compare the middle term anatomic outcomes, complication rates, and operative times of patients with uterovaginal prolapse undergoing VALS with those of women undergoing abdominal sacrocolpopexy.

Methods: This is a prospective cohort study that evaluates operation times, anesthesia times, estimated blood loss, middle term outcomes, perioperative and postoperative complications. We compared the results of 47 women who had the VALS to that of 32 abdominal sacrocolpopexy.

DETAILED DESCRIPTION:
This is a prospective cohort study comparing VALS method to AS with concurrent hysterectomy in patients advanced symptomatic utero vaginal prolapse stage 3 or 4 according to Pelvic Organ Prolapse Quantification (POP-Q) system. This study was carried out from July 2015 to December 2018. Women suffering from prolapse and who desired surgical correction of their prolapse were included to trial. Fertile women who have not completed their family and women with previous POP surgery, POP stage ≤ 2 and women who prefer conservative management or uterus sparing surgery were excluded from the study. Written informed consent was obtained from all patients before enrolment. This study was approved by the institutional review board. Demographic data including age at surgery, parity, menopausal status, body mass index (BMI), previous pelvic surgeries (hysterectomy, pelvic floor repair, etc.), and comorbidities were obtained from the patient's medical records.

Operations:

The VALS procedure consists of two steps. First, vaginal hysterectomy or laparoscopically assisted vaginal hysterectomy performed, anterior vaginal wall dissected up to bladder neck starting from initial vaginal incision, posterior vaginal wall dissected from rectum starting from initial vaginal incision up to distal third of posterior vaginal wall. At this step, eversion of the vaginal walls with the aid of surgeon's fingers would facilitate dissection sharply or bluntly. Two hand-sewn, 15 cm long, 3 cm width type 1 polypropylene meshes transfixed to anterior and posterior vaginal wall with 4-6 polyglactin suture to each wall. The free arms of fixed meshes are introduced to the peritoneal cavity and the vaginal vault is closed with absorbable polyglactin suture. Mid urethral sling and/or perineoplasty were performed vaginally before laparoscopy. After changing gloves of surgery team and setting of endoscopy unit, laparoscopy phase was performed with one intraumbilical (10 mm), 3 lateral abdominal (5 mm) trocars. The sacral promontory is identified and the overlying peritoneum is opened up to vaginal cuff laterally to the rectum and medially to the right uterosacral ligament. Two mesh strips fixated to anterior longitudinal ligament of the sacrum with two separate no: 1 polypropylene sutures without tension. The mesh was then peritonealized with absorbable interrupted extracorporeal sutures.

AS was performed via Pfannenstiel incision after total or subtotal abdominal hysterectomy was performed regarding the surgeon's choice or presence of cervical pathology. Sacrocolpopexy was performed similar to laparoscopic sacrocolpopexy. The rectosigmoid colon was reflected to the left of the midline to expose the presacral area. The sacral promontory is identified and the overlying peritoneum is opened vertically with scissors by sharp dissection up to vaginal cuff laterally to the rectum and medially to the right uterosacral ligament. After placing a sponge stick or sizer to vagina for manipulation and easy identification of dissection plane, anterior vaginal wall dissected from bladder and posterior vaginal wall dissected from rectum. The surgeon has decided the limit of anterior and posterior vaginal wall dissection. The type 1 polyprolene mesh cut and attached with polyprolpelene suture in a Y formation, typically with 5 cm arm length, 3 cm width and 15-18 cm total length. The appropriate length for each patient is determined intraoperatively. The arms of mesh transfixed to anterior and posterior vaginal wall with 4-6 polyglactin suture to each wall starting from distally. Long arm of mesh fixated to anterior longitudinal ligament of the sacrum with two separate no: 1 polypropylene sutures without tension. The excess mesh parts were trimmed over the sacral promontory after the fixation. The mesh was then reperitonealized with absorbable sutures.

We recorded operation times, anesthesia time, additional procedures time, estimated blood loss, outcomes, perioperative and postoperative complications. Anesthesia time began with the anesthetic induction and ended with recovering from anesthesia and transfer of patient to recovery room, including positioning, skin preparation, covering and surgical equipment set up. The total operating time began with the first skin incision and ended with the last closure of an incision. Exclusive operation time of index procedures was calculated by subtracting the additional surgery time from the total operation time.

Early complications were defined as any complication that occurred during surgery or within 4 weeks postoperatively including injury to the bladder, bowel, vagina, ureters, or vessels; wound complications; hematoma, abscess, urinary tract infection, gluteal pain, ileus, blood transfusion, and mesh infection. Late complications described any complications occurred during the entire follow-up period after 4 weeks such as; mesh exposition, mesh extrusion mesh perforation, ileus, dyspareunia, vesicovaginal fistul, rectovaginal fistul, ureter obstruction or fistulization.

Postoperatively, subjects were evaluated for subjective and anatomic outcomes of the operations by vaginal examination at 1 week and 1, 3, and 12months, every years after surgery. Recurrence was defined as stage II or greater apical prolapse, with the leading edge of the C point to 1 cm on either side of the introitus that requires surgical treatment. Objective failure was defined as stage II or greater pelvic organ prolapse, with the leading edge of the prolapse to 1 cm on either side of the introitus. Subjective failure defined as, if the patients responses were "no change" and "minimally/much worse" in Patient Global Impression of Improvement (PGI-I) which used to assess the outcome of surgical treatment [10].

Statistical analysis was performed after normality testing (histogram analysis and/or Kolmogorov-Smirnov testing) using IBM SPSS, version 21 (IBM Inc., Armonk, NY). The student's t-test was used for comparisons of normally distributed variables, the Mann-Whitney U-test was used for non parametric variables, χ2 test and Fisher's exact tests were used to compare categorical variables. A sample size calculation was performed by using data from von Pechman's pilot study assuming that expected difference in means 0.0, standart deviation is 1.3 from LAS study which compares laparoscopic and open sacrocolpopexy [9, 11]. A sample size of 27 for each group was calculated based on these data, 0.05, one-sided t test was estimated to have 80% power to reject the null hypothesis that the VALS and AS techniques are not equivalent.

ELIGIBILITY:
Inclusion Criteria:

- Women suffering from prolapse and who desired surgical correction of their prolapse were included to trial.

Exclusion Criteria:

- Fertile women who have not completed their family and women with previous POP surgery, POP stage ≤ 2 and women who prefer conservative management or uterus sparing surgery were excluded from the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Middle term failure | 2 years
  stage II or greater apical prolapse, with the leading edge of the C point to 1 cm on either side of the introitus that requires surgical treatment

SECONDARY OUTCOMES:
anatomic failure | 2 years
  as stage II or greater pelvic organ prolapse, with the leading edge of the prolapse to 1 cm on either side of the introitus
subjective failure | 2 years
  Subjective failure defined as, if the patients responses were "no change" and "minimally/much worse" in Patient Global Impression of Improvement (PGI-I) which used to assess the outcome of surgical treatment